CLINICAL TRIAL: NCT02708069
Title: e-Unstuck: Interactive e-Learning Software for Parents to Support Executive Functioning and Behavior Regulation in Children With Autism Spectrum Disorder
Brief Title: e-Unstuck:Interactive e-Learning Software for Parents to Support Executive Functioning and Behavior Regulation in Children With Autism Spectrum Disorder
Acronym: e-Unstuck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R44MH109193 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-15 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Autistic Disorder
Keywords: Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Unstuck condition (Other): Parents in the e-Unstuck condition will be asked to complete each of the e-Unstuck modules (one per week) over the course of the nine-week intervention, in addition to reading the UOT manual.
  Interventions: Other: e-Unstuck
- In-Person condition (Other): Parents participating in the in-person condition will be asked to attend two in-person trainings (approximately 125 and 100 minutes respectively) on the Unstuck and On Target (UOT) curriculum, in addition to reading the UOT manual.
  Interventions: Other: Unstuck and On Target

INTERVENTIONS:
Other: e-Unstuck — An e-learning software that delivers the evidence-based Executive Functioning intervention to parents of children with Autism Spectrum Disorder without Intellectual Disability (ASDwoID) with personalized training and feedback on the evidence-based Unstuck and On Target (UOT) curriculum. Through video modeling, intelligent games, adaptive interactive exercises, and personalized feedback, e-Unstuck will provide parents with new tools for applying UOT principles to real world settings, above and beyond learning UOT principles.
  Arms: e-Unstuck condition
Other: Unstuck and On Target — An executive functioning intervention specifically targeted to the needs of the Autism Spectrum Disorder without Intellectual Disability (ASDwoID) population.
  Other Names: UOT
  Arms: In-Person condition

SUMMARY:
The goal of this project is to develop and test e-Unstuck, an e-learning intervention that (1) provides advanced training to parents of children with Autism Spectrum Disorder without Intellectual Disability (ASDwoID) on how to implement the evidence-based Unstuck and On Target (UOT) curriculum at home and (2) is built on 3C's proprietary, state-of-the-art, Dynamic e-Learning Platform, an established platform with high ratings of quality, value, usability, and feasibility from end users. As a result of the pilot efficacy test, the investigators hypothesize that (1) parents who interact with the e-Unstuck software will report greater knowledge and use of UOT principles, less parenting stress and greater parenting sense of competence, and improved child executive function (EF) and social skills compared to control parents, (2) parents who spend more time engaged with the intervention will show greater improvements in outcome variables, and (3) parents who interact with the e-Unstuck software will find the software to be of high quality, value, usability, and feasibility.

DETAILED DESCRIPTION:
Background and Significance: The current prevalence of Autism Spectrum Disorder is 1 in 68 children, and 69% of these children do not have an intellectual disability (ASDwoID). Individuals with ASDwoID are at considerable risk for maladaptive adult outcomes (e.g., un- or underemployment), and executive functioning (EF) impairments significantly contribute to this risk. Unstuck and On Target (UOT) is the only empirically supported EF intervention specifically targeted to the needs of the ASDwoID population. It has improved both EF and social skills in children with ASDwoID in a randomized controlled trial. Despite its demonstrated success, there are significant geographical, scheduling, and financial barriers to parental adaptation of the Unstuck and On Target (UOT) curriculum.

Goal and Innovation: The goal of this project is to develop and test e-Unstuck, an e-learning intervention that (1) provides advanced training to parents of children with ASDwoID on how to implement the evidence-based UOT curriculum at home and (2) is built on 3C's proprietary, state-of-the-art, Dynamic e-Learning Platform, an established platform with high ratings of quality, value, usability, and feasibility from end users. e-Unstuck will make UOT more accessible to parents with geographical, scheduling, and/or financial constraints and will provide parents with key tools (e.g., video modeling, virtual simulations, personalized reports) to increase efficacious adoption of UOT principles, above and beyond those provided in the UOT manual. e-Unstuck will be the first dynamically adaptive, personalized, interactive software product specifically designed to deploy an evidence-based EF intervention to parents of children with ASDwoID.

Specific Aims: The investigators will accomplish five specific aims, two in Phase I, and three in Phase II: (1) develop a prototype of e-Unstuck, (2) conduct a feasibility test of e-Unstuck with parents of children with ASDwoID between the ages of 8-12, (3) fully develop the e-Unstuck software and conduct iterative usability testing with parents of children with ASDwoID, (4) conduct a pilot efficacy test in which 110 parents of children with ASDwoID are randomly assigned to the e-Unstuck intervention or to a control condition in which they receive in-person training on the UOT curriculum, and (5) prepare e-Unstuck for commercialization.

Hypotheses: As a result of the pilot efficacy test, the investigators hypothesize that (1) parents who interact with the e-Unstuck software will report greater knowledge and use of UOT principles, less parenting stress and greater parenting sense of competence, and improved child EF and social skills compared to control parents, (2) parents who spend more time engaged with the intervention will show greater improvements in outcome variables, and (3) parents who interact with the e-Unstuck software will find the software to be of high quality, value, usability, and feasibility.

Commercialization Plan: e-Unstuck will be a unique commercial offering within a large underserved niche market. Revenue will be generated through direct sales to parents of children with ASDwoID and volume sales to organizations (e.g., schools, clinics, parent support agencies) who work with children with ASDwoID and their parents.

ELIGIBILITY:
Inclusion Criteria (Parents):

* be fluent English speakers,
* have a child aged 8-12 years old who has received an ASD diagnosis without intellectual disability from a community mental health professional, and
* have a child that (1) Qualify for an ASD diagnosis based on expert clinical judgment using DSM-5 criteria and by meeting criteria on the Autism Diagnostic Observation Schedule (ADOS), (2) IQ and verbal mental age will not be impaired on an IQ test, and (3) Shift Scale or Plan/Organize Scale will also show clinical impairment on the BRIEF.
* be able to access a computer with internet.
* be able to travel to study sites in Rockville, MD and Washington, DC.

Inclusion Criteria (Children)

* Qualify for an ASD diagnosis based on expert clinical judgment using DSM-5 criteria and Social Affect and Restricted and Repetitive Behavior Total ≥ 7 on the ADOS/ADOS-2,
* IQ ≥ 70 and verbal mental age ≥ 8 years on the WASI-II, and
* Shift Scale or Plan/Organize Scale ≥ 60 on the BRIEF.

Exclusion Criteria:

- Parents who previously participated in feasibility testing (Phase I, Aim 2), usability testing (Phase II, Aim 1), a prior study of the Unstuck and On Target (UOT) curriculum, or in-person training of the UOT curriculum will be excluded due to their familiarity with the curriculum.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ratings of top three child EF difficulties interference with daily functioning as measured on the Top Executive Functioning Difficulties. | After 9 weeks of parental UOT Training
  On this parent-report measure parents rank their child's top 3 EF difficulties and, using a 4 point likert scale (1-no interference to 4-severely interfering), indicate to what extent each difficulty interferes with 5 aspects of their child's daily functioning-daily activities, social activities, follow directions, independence, and task completion. Each difficulty interference score is calculated by summing the 5 rated items and weighted by rank.

SECONDARY OUTCOMES:
Change from baseline in child executive function using the Behavior Rating of Executive Function-II (BRIEF-II). | After 9 weeks of parental UOT Training
  This parent-report questionnaire contains 86 items and assesses child EF skills, including flexibility and planning/organization. For this scale, higher T-scores corresponding to higher levels of executive function impairment.
Change from baseline in parental self-efficacy on the Parenting Sense of Competence Scale. | After 9 weeks of parental UOT Training
  In this 17-item scale, parents report on their satisfaction (e.g., anxiety, motivation) and self-efficacy (e.g., competence, capability) as parents. The index uses a 6 point likert scale (1-strongly agree to 6-strongly disagree). Scoring for multiple items is reverses so that for all items, higher scores indicate greater self-esteem and self-efficacy.
Change from Baseline in parental perceptions of caregiving as measured on the Caregiver Questionnaire | After 9 weeks of parental UOT Training
  This questionnaire contains 21 items and parents report on their sense of child-related strain, competence and empowerment. The items are rated on a 5 point likert scale (1-not at all to 5-very much). Each subscale score is the sum total of the appropriate 7 items, with higher scores indicating higher perceived strain, sense of competence and empowerment.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Childress, PhD, Principal Investigator — 3C Institute; Lauren Kenworthy, PhD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Health System, Rockville, Maryland
  - 3C Institute, Durham, North Carolina